CLINICAL TRIAL: NCT00066664
Title: Characterization of Serum Proteomic Patterns in Neoplastic and Inflammatory Skin Disease
Brief Title: Serum Protein Patterns in Participants With Mycosis Fungoides/Cutaneous T-Cell Lymphoma, Psoriasis, or Normal Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: 030228; 03-C-0228; CDR0000316453; NCT00063167 (obsolete NCT alias)
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Lymphoma
Keywords: recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome

INTERVENTIONS:
Genetic: proteomic profiling

SUMMARY:
RATIONALE: The presence of specific serum proteins may allow a doctor to determine if a patient has mycosis fungoides/cutaneous T-cell lymphoma.

PURPOSE: This clinical trial is studying how well blood protein analysis detects mycosis fungoides/cutaneous T-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether computer-assisted, higher-order analysis of participant low molecular weight serum proteins can detect distinctive proteomic patterns in participants with normal skin vs mycosis fungoides/cutaneous T-cell lymphoma vs psoriasis.
* Determine whether these proteomic patterns can distinguish between various stages of cutaneous T-cell lymphoma.

OUTLINE: This is a pilot study.

Participants complete a general and skin health questionnaire and undergo a whole-body skin examination. Blood samples are taken and analyzed for low molecular weight serum proteins by mass spectroscopy.

PROJECTED ACCRUAL: A total of 141-423 participants (47-94 each of healthy volunteers, psoriasis patients, and T3 cutaneous T-cell lymphoma patients and 141 T1, T2, and T4 mycosis fungoides patients) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets criteria for 1 of the following categories:

  * Healthy skin volunteer

    * No significant inflammatory or neoplastic disease of the skin or internal organs
  * Diagnosis of 1 of the following skin diseases*:

    * Psoriasis

      * Plaque-type disease
      * Psoriasis Area and Severity Index score at least 12
    * Mycosis fungoides/cutaneous T-cell lymphoma

      * Clinical diagnosis of T1-T4 skin disease with a compatible pathologic diagnosis NOTE: *Stable or worsening disease on no therapy or topical therapy only within the past 2 weeks

PATIENT CHARACTERISTICS:

Age

* 18 to 85

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant
* No known HIV-1-related diseases
* No known HTLV-1-related diseases
* Willing to undergo brief skin examination and fill out a questionnaire regarding skin and general health

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 2 weeks since prior systemic therapy for skin disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 423 (Estimated)
Dates: Start 2003-06; Primary Completion 2007-12 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark C. Udey, MD, PhD, Principal Investigator — NCI - Dermatology Branch
Locations (4):
- United States (4):
  - Stanford Cancer Center, Stanford, California
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan

REFERENCES:
- [Background] Liu C, Shea N, Rucker S, Harvey L, Russo P, Saul R, Lopez MF, Mikulskis A, Kuzdzal S, Golenko E, Fishman D, Vonderheid E, Booher S, Cowen EW, Hwang ST, Whiteley GR. Proteomic patterns for classification of ovarian cancer and CTCL serum samples utilizing peak pairs indicative of post-translational modifications. Proteomics. 2007 Nov;7(22):4045-52. doi: 10.1002/pmic.200601044. PMID 17952875
- [Result] Cowen EW, Liu CW, Steinberg SM, Kang S, Vonderheid EC, Kwak HS, Booher S, Petricoin EF, Liotta LA, Whiteley G, Hwang ST. Differentiation of tumour-stage mycosis fungoides, psoriasis vulgaris and normal controls in a pilot study using serum proteomic analysis. Br J Dermatol. 2007 Nov;157(5):946-53. doi: 10.1111/j.1365-2133.2007.08185.x. Epub 2007 Sep 13. PMID 17854367